CLINICAL TRIAL: NCT05450354
Title: Associated Psychiatric Disorders in Children Hospitalized for a Serious Suicide Attempt
Acronym: SuiciDev
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220360; 2022-A00462-41 (Other: ID-RCB Number)
Record Dates: First submitted 2022-06-03; First posted 2022-07-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-10

CONDITIONS: Serious Suicide Attempt
Keywords: Serious suicide attempt in children; Neurodevelopment; Psycho-emotional development; psychopathological characteristics; Attachment disorders; Disorganized attachment
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Alive patients between the ages of 9 and 15 included at the time of their hospitalization at the Necker Enfants Malades Hospital following a serious suicide attempt that took place after January 1, 2016 and at least one of the two parents of the patient, to answer to the study questionnaires.
  Interventions: Other: Questionnaires; Other: Questionnaire
- Control patients: Patients aged 9 to 15 years hospitalized at the Necker-Enfants Malades hospital at time of the study for a non-serious suicide attempt and at least one of the two parents of the patient.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaires — Questionnaires will be completed only once :
  * Neurodevelopment in children: Kiddie Schedule for Affective Disorders and Schizophrenia, Present and Lifetime version (K-SADS-PL-5), the Social Responsiveness Scale (SRS), The Children's Communication Checklist-2 (CCC-2), The Autism-Tics, ADHD and Other Comorbidities Inventory (A-TAC), CONNERS-3, Sensory Profile 2 (DUNN)
  * Psychopathological profile of the child by evaluating the presence of psychotic symptoms: K-SADS-PL-5, Prodromal Questionnaire (F PQ16)
  * Presence of mood and anxiety disorders: Child Depression Inventory (CDI), Revised Children's Manifest Anxiety Scale (RCMAS)
  * Presence of sleep disorders: Children's Sleep Habits Questionnaire (CSHQ). The K-SADS-PL-5 will only be completed by subjects who have attempted suicide after the start of the study; it requires a semi-structured interview of the child by a child psychiatrist and cannot be done remotely. The other scales will be completed by all included subjects.
  Groups: Patients
Other: Questionnaire — Determination of attachment style : Adolescent Relationship Scale Questionnaire (ARSQ). The questionnaire will be completed only once.

SUMMARY:
Several studies agree on the increase in suicide attempts in children over the past 15 years. This trend has been aggravated by the COVID 19 pandemic.

It is recognized that suicide attempts are mostly encountered in individuals with a psychiatric disorder. Serious suicide attempts, which probably better reflect the risk of completed suicide, are very poorly known and have been very little explored. They could be related to more specific and earlier psychiatric disorders or even concern children with developmental particularities that are insufficiently defined to fall under a categorical diagnosis, but which could be better understood with dimensional measurements. Better characterizing them would seem quite important given their high lethality. Indeed, a high lethality is found for half of the suicide attempts in children fewer than 12, contrasting with a moderate or low intentionality ; in children, the means used are often more violent and more lethal than in adolescents (over 12 years old): hanging, firearm, etc.

The Necker-Enfants Malades hospital has a pediatric neurosurgery department as well as a specialized multidisciplinary team to care for polytraumatized children in a regional "Trauma Center" type structure. As a result, most children and adolescents in Ile-de-France who have made a violent suicide attempt are sent to the Necker hospital. Once medico-surgically stabilized, these children and adolescents are assessed by the hospital's child psychiatry team. This regional recruitment makes it possible to have an epidemiological representativeness. From this population, the investigative team proposes to better characterize the developmental profile and psychiatric disorders of children who have made a serious suicide attempt.

The study also proposes to examine in detail the psycho-emotional development as well as the psychopathological characteristics of these children in order to shed light on these early and lethal acting out. The investigative team proposes in particular to use dimensional evaluations to analyze behavioral traits in more detail. To the knowledge of the child psychiatry department of the Necker Enfants Malades hospital, there is no such study to date.

In addition to the question of neurodevelopmental disorders, an ancillary study will make it possible to question attachment disorders in children who have made a serious suicide attempt.

In fact, a link between attachment disorders and suicidal ideation or attempted suicide has been shown in the literature.

Attachment disorders correspond to an early imbalance in the bond between a child and the primary caregiver, particularly before the age of 3. Attachment relationships that do not allow a solid bond between the young child and the person occupying the maternal function may not be pathological in themselves but would be risk factors for pathologies in adolescence and adulthood, and in particular a category of so-called disorganized attachment disorders in the occurrence of dissociative symptoms.

DETAILED DESCRIPTION:
In 2016, the French national institute of statistics and economic studies (INSEE) indicates about the death of children aged 5 to 14 in France, that 4.2% of deaths at this age (n=26) are due to suicide, with a possible sub- assessment of suicide in this age group because a certain number of deaths are attributed to accidents.

Several studies agree on the increase in suicide attempts in children over the past 15 years. This trend has been aggravated by the COVID 19 pandemic. Indeed, several recent studies have reported deterioration in the mental health of children and adolescents since the start of the pandemic and an increase in the rate of suicidal ideation and suicide attempts in 2020. Among the factors that could explain this increase, we can cite the phenomena of social distancing and isolation.

It is recognized that suicide attempts are mostly encountered in individuals with a psychiatric disorder. Indeed, psychological autopsies indicate a prevalence of psychiatric disorders of more than 90% among people who died by suicide.

Nevertheless, serious suicide attempts, which probably better reflect the risk of completed suicide, are very poorly known and have been very little explored. They could be related to more specific and earlier psychiatric disorders or even concern children with developmental particularities that are insufficiently defined to fall under a categorical diagnosis, but which could be better understood with dimensional measurements. Better characterizing them would seem quite important given their high lethality. Indeed, a high lethality is found for half of the suicide attempts in children fewer than 12, contrasting with a moderate or low intentionality ; in children, the means used are often more violent and more lethal than in adolescents (over 12 years old): hanging, firearm, etc.

The Necker-Enfants Malades hospital has a pediatric neurosurgery department as well as a specialized multidisciplinary team to care for polytraumatized children in a regional "Trauma Center" type structure. As a result, most children and adolescents in Ile-de-France who have made a violent suicide attempt are sent to the Necker hospital. Once medico-surgically stabilized, these children and adolescents are assessed by the hospital's child psychiatry team. This regional recruitment makes it possible to have an epidemiological representativeness. From this population, the investigative team proposes to better characterize the developmental profile and psychiatric disorders of children who have made a serious suicide attempt.

The study also proposes to examine in detail the psycho-emotional development as well as the psychopathological characteristics of these children in order to shed light on these early and lethal acting out. The investigative team proposes in particular to use dimensional evaluations to analyze behavioral traits in more detail. To the knowledge of the child psychiatry department of the Necker Enfants Malades hospital, there is no such study to date.

In addition to the question of neurodevelopmental disorders, an ancillary study will make it possible to question attachment disorders in children who have made a serious suicide attempt.

In fact, a link between attachment disorders and suicidal ideation or attempted suicide has been shown in the literature.

Attachment disorders correspond to an early imbalance in the bond between a child and the primary caregiver, particularly before the age of 3. Attachment relationships that do not allow a solid bond between the young child and the person occupying the maternal function may not be pathological in themselves but would be risk factors for pathologies in adolescence and adulthood, and in particular a category of so-called disorganized attachment disorders in the occurrence of dissociative symptoms.

The adolescent relationship scale questionnaire (ARSQ), to determine attachment style, will be offered to children and adolescents who have made serious suicide attempts who will participate in the study as well as to a control group of children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Between the ages of 9 and 15 inclusive at the time of hospitalization at the Necker Enfants Malades Hospital following a serious suicide attempt that took place after January 1, 2016.
  * Serious suicide attempt whose criteria are: hospitalization for more than 24 hours and one of the following criteria: care in a specialized service, surgery under general anesthesia, hospitalization in intensive care or continuous care or resuscitation unit, attempted suicide by methods involving a high risk of mortality: precipitation, hanging, firearm…
  * Control patients aged 9 to 15 years old hospitalized at the Necker-Enfants Malades hospital at time of the study for a non-serious suicide attempt.
  * Without intellectual disability (IQ>70).
* Parents:

  - At least one of the parents of a patient meeting the inclusion criteria.
* All subjects (parent(s) and minor or adult children) informed and not objecting to participation in the study. Holders of parental authority of minor patients informed and not opposing the participation of their child in the study.

Exclusion Criteria:

* Insufficient command of French to answer the questionnaires.
* Incomplete file of patients whose hospitalization is no longer in progress.
* Medical impossibility to pass the questionnaires.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Alive patients who made a serious suicide attempt between the ages of 9 and 15 inclusive and after January 1, 2016. And control patients aged 9 to 15 years old hospitalized at the Necker-Enfants Malades hospital at time of the study for a non-serious suicide attempt.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Description of the distribution of scores of the Autism-Tics, ADHD and Other Comorbidities Inventory (A-TAC) assessing neurodevelopment | Day 0
  A-TAC is a hetero-questionnaire of 96 "gate items" used for basic screening and identification of proxies to diagnoses, organized in different modules, and 163 additional items tapping into more specific symptoms including 72 items (4/module) addressing psychosocial dysfunction and subjective suffering associated with that particular problem area, the age at onset and whether the problems are present or in remission. 3 answers are possible/item (yes, scored 1; yes to some extent, 0,5; no, 0). For each module in which at least one item is answered in the affirmative, the parents tell about whether or not the endorsed symptoms had led to (1) dysfunction at school, among peers, or at home, and (2) suffering on the part of the child. A "problem load score" is calculated as the sum of these 2 items (from 0 to 2), with a theoretically defined cut-off for problems "significant" at ≥ 1, indicating that one of the problem questions is fully endorsed or that both are endorsed "to some extent".

SECONDARY OUTCOMES:
Evaluation of neurodevelopment by a dimensional scale (K-SADS-PL-5) | Day 0
  Kiddie Schedule for Affective Disorders and Schizophrenia, Present and Lifetime version (K-SADS-PL-5) : Semi-structured diagnostic interview to assess mental disorders in children and adolescents (6-18 years). It includes a dimensional and categorical assessment of the symptoms of current and past episodes of psychopathology, in order to make one or more diagnoses according to the DSM-5 criteria. For each category related to DMS-5 diagnosis, there are 4 possible answers for the most severe past episode (0: no information; 1: no diagnosis; 2: likely diagnosis, 3: clear diagnosis) and 5 possible answers for the actual episode (0: no information; 1: no diagnosis; 2: likely diagnosis, 3: clear diagnosis; 4: in partial remission).
Evaluation of neurodevelopment by a dimensional scale (SRS) | Day 0
  Social Responsiveness Scale (SRS) : 65-item hetero-questionnaires for children and adolescents from 4 to 18 years old concerning social awareness, cognition, communication and motivation, repetitive behaviors and restricted interests. Each item on the scale inquires about an observed aspect of reciprocal social behaviour that is rated on a scale from "0" (never true) to "3" (almost always true).
Evaluation of neurodevelopment by a dimensional scale (CCC-2) | Day 0
  Children's Communication Checklist (CCC-2) : 70-item hetero-questionnaire for children and adolescents from 4 to 16 years old which evaluates the structure of language, pragmatic difficulties and non-linguistic aspects of autistic behaviors (social relations and centers of interest). It does not allow the diagnosis of autism spectrum disorder. It quantifies the strengths and weaknesses of children's communication from 0 ("less than once a week") to 3 ("every day").
Evaluation of neurodevelopment by a dimensional scale (CONNERS-3) | Day 0
  CONNERS-3 : 108-item hetero-questionnaire to assess the presence of symptoms of inattention, hyperactivity, impulsivity and other frequently associated disorders in children and adolescents aged 6 to 18. Symptoms are rated on a Likert scale with severity ratings from 0 (not at all/never) to 3 (very much/ very frequently).
Evaluation of neurodevelopment by a dimensional scale (DUNN) | Day 0
  Sensory Profile 2 (DUNN) : hetero-questionnaire of 86 items evaluating the behavioral reactions of the child in response to sensory stimuli as well as their repercussions on occupational performance in children and adolescents from 3 to 15 years old. There are 5 possible answers for each item (always, scored as 1; frequently, scored as 2; sometimes, scored as 3; rarely scored as 4; and never scored as 5).
Correlation between neurodevelopmental particularities and the age of suicide attempt | Day 0
  Study of the correlation between the presence of neurodevelopmental particularities assessed by the dimensional scales (K-SADS-PL-5, A-TAC, SRS, CCC-2, CONNERS-3, DUNN) and the age of suicide attempt.
Presence of psychotic symptoms | Day 0
  Description of scale scores to assess the presence of psychotic symptoms in children who have made a serious suicide attempt.
  Prodromal Questionnaire French Version (F PQ16) : self-administered 16-item questionnaire for individuals under 35 years of age assessing the presence of attenuated psychotic symptoms. The cut-off for a significant presence of psychotic symptoms is ≥ 4 of the 16 items.
Description of associated mood disorders in children who have made a serious suicide attempt | Day 0
  Child Depression Inventory (CDI) : Self-questionnaire of 27 items which measures the intensity of depression in children and adolescents from 7 to 17 years old. Each item is rated from 0 (normal behavior for age or absent) to 2 (severe). The addition of the items gives a total between 0 and 54. The higher the score, the more severe the depression symptomatology is.
  Revised Children's Manifest Anxiety Scale (RCMAS) : Self-administered 37-item questionnaire assessing the level and nature of anxiety in children and adolescents aged 9 to 19, not allowing diagnosis of the various anxiety disorders in children. The total anxiety score can range from 0 to 28. The cut-off point for pathological anxiety is more than two standard deviations around the mean (T>70).
Description of sleep characteristics in children who have made a serious suicide attempt | Day 0
  Children's Sleep Habits Questionnaire (CSHQ): 33-items hetero-questionnaire to assess sleep habits in children aged 4 to 10, validated in adolescents up to 17 years old. There are 3 possible answers for each item (rarely, scored as 1; sometimes, scored as 2; and regularly scored as 3).
Description of the distribution of scores of the Adolescent Relationship Scale Questionnaire (ARSQ) assessing the style of attachment | Day 0
  Self-questionnaire of 17 items rated 1 = Not at all like me, at 5=Totally like me, allowing to distinguish the 4 different attachment styles (secure, preoccupied, ambivalent, disorganized). The results of patients who made a serious suicide attempt will be compared with those of patients who made non-serious suicide attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Mélisande Sansen, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Pauline Chaste, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy-Bencheton J, Chaste P, Sansen M. Link between neurodevelopmental disorders and suicidal risk in children. Encephale. 2025 Feb;51(1):39-45. doi: 10.1016/j.encep.2023.12.002. Epub 2024 Mar 23. PMID 38523026
- [Background] Skovgaard AM. Mental health problems and psychopathology in infancy and early childhood. An epidemiological study. Dan Med Bull. 2010 Oct;57(10):B4193. PMID 21040689
- [Background] https://www.who.int/fr/news-room/fact-sheets/detail/suicide
- [Background] Stordeur C, Acquaviva E, Galdon L, Mercier JC, Titomanlio L, Delorme R. [Suicide attempts in children under 12 years of age]. Arch Pediatr. 2015 Mar;22(3):255-9. doi: 10.1016/j.arcped.2014.12.004. Epub 2015 Feb 2. French. PMID 25656458
- [Background] Scharfe E., Reliability and Validity of an Interview Assessment of Attachment Representations in a Clinical Sample of Adolescents 2002
- [Background] Rosen DH. The serious suicide attempt. Five-year follow-up study of 886 patients. JAMA. 1976 May 10;235(19):2105-9. doi: 10.1001/jama.235.19.2105. PMID 946536
- [Background] Prior V, Glaser D. Comprendre l'attachement et les troubles de l'attachement : théorie, preuve et pratique. Bruxelles : De Boeck ; 2010
- [Background] National Center for Injury Prevention and Control-blank template
- [Background] Lyons-Ruth K, Dutra L, Schuder MR, Bianchi I. From infant attachment disorganization to adult dissociation: relational adaptations or traumatic experiences? Psychiatr Clin North Am. 2006 Mar;29(1):63-86, viii. doi: 10.1016/j.psc.2005.10.011. No abstract available. PMID 16530587
- [Background] Liotti G. A model of dissociation based on attachment theory and research. J Trauma Dissociation. 2006;7(4):55-73. doi: 10.1300/J229v07n04_04. PMID 17182493
- [Background] Liotti G. Disorganized/disoriented attachment in the etiology of the dissociative disorders. Dissociation 1992
- [Background] Levi-Belz Y, Beautrais A. Serious Suicide Attempts. Crisis. 2016 Jul;37(4):299-309. doi: 10.1027/0227-5910/a000386. Epub 2016 Jun 1. PMID 27245812
- [Background] Leary MR, Hoyle RH, éditeurs. Handbook of individual differences in social behavior. New York: Guilford Press; 2009
- [Background] Hesse E, Main M. Disorganized infant, child, and adult attachment: collapse in behavioral and attentional strategies. J Am Psychoanal Assoc. 2000;48(4):1097-127; discussion 1175-87. doi: 10.1177/00030651000480041101. PMID 11212184
- [Background] Guedeney N, Fermanian J, Bifulco A. [Construct validation study of the Relationship Scales Questionnaire (RSQ) on an adult sample]. Encephale. 2010 Feb;36(1):69-76. doi: 10.1016/j.encep.2008.12.006. Epub 2009 Apr 7. French. PMID 20159199
- [Background] Guédeney N., S. Tereno b, J. Tissier c, A. Guédeney d, T. Greacen e, T. Saïas e, F. Tubach c, R. Dugravier f, B. Welniarz g , Groupe CAPEDP-A Transmission du traumatisme. La question de l'attachement désorganisé : de la théorie à la pratique ; 2012
- [Background] Guédeney N, Guédeney A, Fonagy P. L'attachement : approche théorique : du bébé́ à la personne âgée: Elsevier Masson ; 2016
- [Background] Conversy L, A Guedeney , Les trouble de l'attachement ; 2017
- [Background] Beautrais AL. Suicide and serious suicide attempts in youth: a multiple-group comparison study. Am J Psychiatry. 2003 Jun;160(6):1093-9. doi: 10.1176/appi.ajp.160.6.1093. PMID 12777267
- [Background] Boris NW, Zeanah CH. Disturbances and disorders of attachment in infancy: an overview. Infant mental health journal 1999
- [Background] Barach PM. Multiple personality disorder as an attachment disorder. Dissociation 1991
- [Background] Ainsworth M, Patterns of attachment : a psychological study on the strange situation, 1978